CLINICAL TRIAL: NCT00176813
Title: Phase II Study of Gemcitabine, Cisplatin, and Celecoxib in the Treatment of Metastatic Pancreatic Cancer
Brief Title: Gemcitabine, Cisplatin, and Celecoxib Treatment of Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Dr. Mark Zalupski, University of Michigan Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2001-071; C2442
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin; Celecoxib

INTERVENTIONS:
Drug: Gemcitabine
Drug: Cisplatin
Drug: Celecoxib

SUMMARY:
This study will examine an investigational (experimental) treatment using gemcitabine, cisplatin, and celecoxib. Preliminary studies have shown that this experimental treatment may be effective in reducing the size of cancerous tumors and/or preventing further tumor growth.

This is a phase II clinical trial studying the reactions of the patient's body and their tumor to the combination of gemcitabine, cisplatin, and celecoxib. The purpose of this study is to see if the tumor responds to this treatment and to determine how long the response lasts. This study will also look at what kind of side effects this experimental treatment causes and see how often these side effects occur. Blood levels of celecoxib will be measured to find out how this treatment affects factors (proteins) involved in new blood vessel formation and tumor growth (angiogenesis).

ELIGIBILITY:
Inclusion Criteria

1. Patients must have histologic or cytologic diagnosis of pancreatic adenocarcinoma.
2. Patients must have clinical/radiologic evidence of metastatic disease (stage IV).
3. Patients must not have received prior chemotherapy for metastatic disease. Prior adjuvant chemotherapy is allowed, provided that the last day of therapy was at least 6 months prior to starting treatment.
4. Patients must have performance status of 0-2 on the SWOG scale.
5. Patients must have an estimated life expectancy of at least 12 weeks.
6. Patients must have adequate bone marrow function: absolute neutrophil count >1,500/cmm, platelet count >100,000/cmm.
7. Patients must be informed of the investigational nature of this study and must give written informed consent prior to the receiving of treatment per this protocol.
8. Patients must practice effective birth control while receiving treatment.

Exclusion Criteria

1. Patients with endocrine tumors or lymphoma of the pancreas.
2. Patients with locally advanced pancreatic cancer.
3. Patients with a proven history (radiographic and/or endoscopic) of peptic ulcer or esophageal erosions within one year of enrollment onto the study.
4. Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other non-steroidal anti-inflammatory drugs.
5. History of active central nervous system (CNS) metastases.
6. Inadequate liver function (bilirubin >3.0 mg/dL); transaminases (AST/ALT) >3 times upper limit of institutional normal.
7. Inadequate renal function (creatinine >1.5 mg/dL).
8. Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
9. History of other malignancy, except for cancers that have been treated with a curative intent and patient is without evidence of active disease.
10. Unresolved bacterial infection requiring treatment with antibiotics.
11. Pregnant or lactating women may not participate in the study.
12. Patients who have allergy to any of the study drugs or sulfa drugs.
13. Patients infected with HIV-1 virus because of the undetermined effect of this chemotherapy regimen in patients with HIV-1 and the potential for serious interaction with anti-HIV medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-03; Primary Completion 2003-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To determine the overall survival time in patients with metastatic pancreatic cancer treated with the combination of gemcitabine, cisplatin and celecoxib. | 12 months

SECONDARY OUTCOMES:
To obtain data on overall time to disease progression | 12 months
To determine time to treatment failure | 12 months
To determine the tolerability of celecoxib with gemcitabine and cisplatin. | 12 months
To characterize the nature of the toxicity for this combination in this patient group. | 12 months
To determine objective tumor response | 12 months
To determine the influence of therapy on the blood levels of prostaglandins and angiogenesis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States